CLINICAL TRIAL: NCT03631381
Title: Retrospective Study of Carotid Surgery in Dijon
Acronym: RESCADI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: STEINMETZ 2017
Record Dates: First submitted 2018-08-10; First posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Carotid Stenosis
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The results in carotid surgery are an indicator of the functioning of an academic surgical team, making it possible to evaluate and improve practices, as much among surgeons in training as among senior surgeons.

The indications have evolved with the development of symptomatic stenosis surgery, and results analysis has allowed us to improve our practices.

It would be of great use to have the statistics obtained in previous years to continue improving our practices.

ELIGIBILITY:
Inclusion Criteria:

all patients operated for carotid stenosis at Dijon University Hospital

Exclusion Criteria:

none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients operated for carotid stenosis in the cardiovascular and thoracic surgery department at Dijon University Hospital since 2000
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-09-04 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
mortality rate (%) | Day 30
incidence of complications (%) | Day 30

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France